CLINICAL TRIAL: NCT01172561
Title: Reducing Cervical Cancer in Appalachia
Brief Title: Community Awareness Resources and Education - Project 1
Acronym: CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Electra Paskett, Professor, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: OSU-0488; P50CA105632 (NIH); NCI-2012-00212 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care Group (Active Comparator): All women over age 18 encouraged to obtain Pap smears appropriate for their risk profile, the comparison arm included a low-literacy brochure to encourage women to receive screening. The brochure was designed to answer basic questions about Pap smears and provide instructions on how to obtain a Pap smear.
  Interventions: Behavioral: Usual Care Group
- Lay Health Advisor Intervention (Experimental): The Lay Health Advisor education intervention - The intervention consisted of an intensive, reinforced, one on one, interactive ed. program (an initial meeting, then 2 calls and a series of 4 postcards mailed at regular intervals and a 2nd visit. Woman were enrolled for about 12 to 14 months.
  Interventions: Behavioral: Lay Health Advisor Education Intervention

INTERVENTIONS:
Behavioral: Lay Health Advisor Education Intervention — The individualized health education intervention consisted of an intensive, reinforced, face to face, interactive educational program. The program included an initial meeting of 45 60 minutes, followed by two telephone calls and reinforcement by a series of four postcards mailed at regular intervals and a second visit. Each woman will be enrolled in the intervention program for approximately 12 to 14 months.
  Arms: Lay Health Advisor Intervention
Behavioral: Usual Care Group — All women over age 18 encouraged to obtain Pap smears appropriate for their risk profile, the comparison arm included a low-literacy brochure to encourage women to receive screening. The brochure was designed to answer basic questions about Pap smears and provide instructions on how to obtain a Pap smear.
  Arms: Usual Care Group

SUMMARY:
To increase early detection of cervical cancer by increasing the proportion of Appalachian women, age 18 and older, who receive Pap smears at appropriate intervals and return for follow-up care when necessary.

DETAILED DESCRIPTION:
The overall goal of Project 1 is to increase early detection of cervical cancer by increasing the proportion of Appalachian women, age 18 and older, who receive Pap smears at appropriate intervals and return for follow-up care when necessary. The project was implemented in Appalachian Ohio, a mainly rural and underserved area with a population comprised of 1.5 million adults, aged 18 and older, and used community-based participatory research (CBPR) and community relationships already established in the area by Center investigators.

ELIGIBILITY:
Inclusion Criteria:

* women age 18 and older

  * who have visited participating clinics during the last two years and
  * who consider themselves to be a current patient of that clinic

Exclusion Criteria:

* Not a resident of the selected Ohio Appalachia county
* Under the age of 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2005-03-01 (Actual); Primary Completion 2008-05-31 (Actual); Study Completion 2009-03-31 (Actual)

PRIMARY OUTCOMES:
Receipt of Cervical Cancer screening via Pap Test | past 12-14 months (yes/no).
  the primary outcome of interest for Project 1 intervention will be a dichotomous variable, Pap smear in the past 12-14 months (yes/no). Initially, We will assess the univariate difference between treatment groups (lay health advisor vs. brochure and physician letter) in the proportion of women who received a Pap smear during the past 12 months using design-based logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Electra D Paskett, Ph.D., Principal Investigator — The Ohio State University Comprehensive Cancer Center
Locations (1):
- The Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paskett ED, McLaughlin JM, Lehman AM, Katz ML, Tatum CM, Oliveri JM. Evaluating the efficacy of lay health advisors for increasing risk-appropriate Pap test screening: a randomized controlled trial among Ohio Appalachian women. Cancer Epidemiol Biomarkers Prev. 2011 May;20(5):835-43. doi: 10.1158/1055-9965.EPI-10-0880. Epub 2011 Mar 23. PMID 21430302
- See also: Jamesline — http://cancer.osu.edu